CLINICAL TRIAL: NCT02493855
Title: An Exploratory Study to Evaluate the Kinetics of Viral Load Decline With Ombitasvir/ABT 450/Ritonavir (Ombitasvir/ABT-450/r) and Dasabuvir Therapy With Low Dose Ribavirin (RBV), Full Dose RBV or RBV Add-On in Treatment Naïve Adults With Genotype 1a Chronic Hepatitis C Virus (HCV) Infection
Brief Title: Ombitasvir/ABT-450/Ritonavir and Dasabuvir Therapy With Low Dose Ribavirin (RBV), Full Dose RBV or RBV Add-On in Treatment Naive Genotype 1a Hepatitis C Virus Infected Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M14-242; 2014-001478-32 (EudraCT Number)
Record Dates: First submitted 2015-07-02; First posted 2015-07-10 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-09

CONDITIONS: Chronic Hepatitis C; Hepatitis C (HCV); Hepatitis C Genotype 1a
Keywords: Treatment naive; HCV; Interferon free; Hepatitis C Genotype 1a; Chronic Hepatitis C; Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — dasabuvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A: Ribavirin Full Dose for Last 10 Weeks (Experimental): Participants received ombitasvir/ABT-450/ritonavir 25 mg/150 mg/100 mg once daily (QD) + dasabuvir 250 mg twice daily (BID) for 12 weeks and weight-based ribavirin (1000 mg or 1200 mg split BID) for the last 10 weeks.
  Interventions: Drug: Ombitasvir/ABT-450/Ritonavir; Drug: Dasabuvir; Drug: Ribavirin (RBV)
- Arm B: Ribavirin Full Dose for 12 Weeks (Experimental): Participants received ombitasvir/ABT-450/ritonavir 25 mg/150 mg/100 mg once daily (QD) + dasabuvir 250 mg twice daily (BID) and weight-based ribavirin (1000 mg or 1200 mg split BID) for 12 weeks.
  Interventions: Drug: Ombitasvir/ABT-450/Ritonavir; Drug: Dasabuvir; Drug: Ribavirin (RBV)
- Arm C: Ribavirin Low-dose for 12 Weeks (Experimental): Participants received ombitasvir/ABT-450/ritonavir 25 mg/150 mg/100 mg once daily (QD) + dasabuvir 250 mg twice daily (BID) and 600 mg ribavirin once daily for 12 weeks.
  Interventions: Drug: Ombitasvir/ABT-450/Ritonavir; Drug: Dasabuvir; Drug: Ribavirin (RBV)

INTERVENTIONS:
Drug: Ombitasvir/ABT-450/Ritonavir — Ombitasvir/ABT-450/ritonavir combination tablets
  Other Names: ABT-267/ABT-450/ritonavir
Drug: Dasabuvir — Dasabuvir tablets
  Other Names: ABT-333
Drug: Ribavirin (RBV) — Ribavirin tablets

SUMMARY:
To evaluate the effect of ribavirin on second phase plasma hepatitis C virus (HCV) ribonucleic acid (RNA) decline in participants who receive ombitasvir/ABT-450/ritonavir and dasabuvir with full dose ribavirin, low dose ribavirin or without ribavirin for 2 weeks in treatment-naive HCV genotype (GT) 1a-infected adults.

ELIGIBILITY:
Inclusion Criteria:

1. Screening laboratory result indicating HCV genotype 1 (GT1) a infection.
2. Chronic HCV infection.
3. Subjects must be non-cirrhotic.
4. Subjects must be able to understand and adhere to the study visit schedule and all protocol requirements as well as voluntarily sign and date an institutional review board (IRB) approved informed consent.

Exclusion Criteria:

1. Women who are pregnant or breastfeeding.
2. Positive test result for hepatitis B surface antigen (HBsAg) or anti-human immunodeficiency virus antibody (HIV Ab) positive immunoassay.
3. Clinically significant abnormalities or co-morbidities, other than HCV infection, that make the subject unsuitable for this study or treatment.
4. Current enrollment in another interventional clinical study. Previous use of any HCV treatments including pegylated interferon (pegIFN), ribavirin, or any direct acting antiviral agent, either investigational or approved, for HCV including protease inhibitors, nucleoside or non-nucleoside polymerase inhibitors, or nonstructural viral protein 5A (NS5A) inhibitors.
5. History or solid organ transplant.
6. Screening laboratory analysis that shows abnormal results.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Dumas, PhD, Study Director — AbbVie

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at one clinic in France and one clinic in the United States. Participants were treatment-naïve adults with hepatitis C virus (HCV) genotype (GT)1a infection without cirrhosis.
Pre-assignment Details: Participants were randomized to Arms A or B in a 1:1 ratio first, and once those arms fully enrolled, Arm C was enrolled. Randomization to Arms A and B was stratified by site.
Period: Overall Study
Arm/Group | Arm A: Ribavirin Full Dose for Last 10 Weeks | Arm B: Ribavirin Full Dose for 12 Weeks | Arm C: Ribavirin Low-dose for 12 Weeks
Started | 21 | 19 | 6
Completed | 19 | 18 | 6
Not Completed | 2 | 1 | 0
Not completed — Non-compliance | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Ribavirin Full Dose for Last 10 Weeks | Arm B: Ribavirin Full Dose for 12 Weeks | Arm C: Ribavirin Low-dose for 12 Weeks | Total
Number analyzed (Participants) | 21 | 19 | 6 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (11.96) | 46.0 (12.78) | 36.7 (15.79) | 44.3 (12.88)
Age, Customized [Count of Participants; unit: Participants]
  < 55 years | 17 | 14 | 5 | 36
  ≥ 55 - 65 years | 4 | 5 | 1 | 10
  ≥ 65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 4 | 27
  Male | 10 | 7 | 2 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 16 | 14 | 4 | 34
  Black of African American | 4 | 3 | 1 | 8
  Asian | 0 | 0 | 0 | 0
  American Indian or Alaskan Native | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Mutli Race | 1 | 2 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Slope of the Second Phase Decline in Plasma HCV Ribonucleic Acid (RNA) Levels During Treatment
Description: HCV viral kinetics in plasma during therapy were modeled through non-linear mixed effect models, including a rapid first phase of initial decline and a slower second phase decline. The slope of the second phase decline was estimated for each treatment arm.
Time Frame: From Week 0 to Week 2
Population: Participants with evaluable HCV RNA to calculate the slope of the second phase. Three participants were excluded due to algorithm non-convergence in the non-linear modeling process.
Measure: Median (Full Range); unit: 1/day
Arm/Group | Arm A: Ribavirin Full Dose for Last 10 Weeks | Arm B: Ribavirin Full Dose for 12 Weeks | Arm C: Ribavirin Low-dose for 12 Weeks
Number analyzed (Participants) | 20 | 17 | 6
1/day | 0.0036 [0.0006 to 0.0128] | 0.0046 [-0.0003 to 0.0155] | 0.0051 [0.0031 to 0.0076]
Statistical Analysis 1: Comparison: Arm A: Ribavirin Full Dose for Last 10 Weeks vs Arm B: Ribavirin Full Dose for 12 Weeks; Test type: Superiority — This study was an exploratory study to evaluate the effect of ribavirin on the slope of the second phase of HCV RNA decline in participants who received the 3-direct-acting antiviral agent regimen; p = 0.311, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Arm B: Ribavirin Full Dose for 12 Weeks vs Arm C: Ribavirin Low-dose for 12 Weeks; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.561, Wilcoxon Rank Sum Test

ADVERSE EVENTS:
Time Frame: From first dose of study drug until 30 days after last dose; up to 16 weeks.
Arm/Group | Arm A: Ribavirin Full Dose for Last 10 Weeks | Arm B: Ribavirin Full Dose for 12 Weeks | Arm C: Ribavirin Low-dose for 12 Weeks
Serious Adverse Events (participants affected / at risk) | 1/21 | 0/19 | 0/6
Other Adverse Events (participants affected / at risk) | 17/21 | 16/19 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Ribavirin Full Dose for Last 10 Weeks (N=21) | Arm B: Ribavirin Full Dose for 12 Weeks (N=19) | Arm C: Ribavirin Low-dose for 12 Weeks (N=6)
DEPRESSION (Psychiatric disorders) | 1 | 0 | 0
DRUG DEPENDENCE (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Ribavirin Full Dose for Last 10 Weeks (N=21) | Arm B: Ribavirin Full Dose for 12 Weeks (N=19) | Arm C: Ribavirin Low-dose for 12 Weeks (N=6)
ANAEMIA (Blood and lymphatic system disorders) | 4 | 4 | 2
INCREASED TENDENCY TO BRUISE (Blood and lymphatic system disorders) | 0 | 1 | 0
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 | 1 | 0
PALPITATIONS (Cardiac disorders) | 0 | 1 | 0
VERTIGO (Ear and labyrinth disorders) | 0 | 2 | 0
DRY EYE (Eye disorders) | 0 | 0 | 1
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 | 3 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 2 | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 1 | 0 | 1
DRY MOUTH (Gastrointestinal disorders) | 1 | 1 | 2
DYSPEPSIA (Gastrointestinal disorders) | 0 | 2 | 3
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 | 0 | 1
NAUSEA (Gastrointestinal disorders) | 3 | 3 | 2
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0
VOMITING (Gastrointestinal disorders) | 3 | 0 | 1
ASTHENIA (General disorders) | 3 | 3 | 0
FATIGUE (General disorders) | 5 | 7 | 2
FEELING ABNORMAL (General disorders) | 0 | 1 | 0
PYREXIA (General disorders) | 0 | 0 | 1
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 2 | 0 | 2
HYPERTRANSAMINASAEMIA (Hepatobiliary disorders) | 0 | 1 | 0
BRONCHITIS (Infections and infestations) | 0 | 1 | 0
FUNGAL SKIN INFECTION (Infections and infestations) | 0 | 1 | 0
INFLUENZA (Infections and infestations) | 1 | 0 | 0
ORAL CANDIDIASIS (Infections and infestations) | 0 | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0 | 1
LIMB INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 1
PROCEDURAL HEADACHE (Injury, poisoning and procedural complications) | 0 | 1 | 0
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 7 | 5 | 5
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 0 | 1 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1 | 0
BODY TEMPERATURE FLUCTUATION (Investigations) | 0 | 0 | 1
GLUCOSE URINE PRESENT (Investigations) | 0 | 1 | 0
HAEMOGLOBIN DECREASED (Investigations) | 1 | 3 | 0
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 0 | 1 | 0
PROTHROMBIN LEVEL INCREASED (Investigations) | 0 | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 0 | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0
HYPERMAGNESAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
MUSCLE TIGHTNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
AMNESIA (Nervous system disorders) | 0 | 1 | 0
DIZZINESS (Nervous system disorders) | 0 | 2 | 0
HEADACHE (Nervous system disorders) | 4 | 4 | 0
MEMORY IMPAIRMENT (Nervous system disorders) | 0 | 3 | 0
MIGRAINE (Nervous system disorders) | 0 | 1 | 0
SYNCOPE (Nervous system disorders) | 1 | 1 | 0
ANXIETY (Psychiatric disorders) | 1 | 0 | 1
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 0 | 1
DEPRESSED MOOD (Psychiatric disorders) | 0 | 1 | 0
DEPRESSION (Psychiatric disorders) | 3 | 2 | 0
EMOTIONAL DISTRESS (Psychiatric disorders) | 0 | 1 | 0
INSOMNIA (Psychiatric disorders) | 3 | 3 | 0
IRRITABILITY (Psychiatric disorders) | 0 | 1 | 0
MOOD SWINGS (Psychiatric disorders) | 0 | 0 | 1
SLEEP DISORDER (Psychiatric disorders) | 0 | 0 | 1
CHROMATURIA (Renal and urinary disorders) | 0 | 1 | 0
DYSURIA (Renal and urinary disorders) | 0 | 0 | 1
POLYMENORRHOEA (Reproductive system and breast disorders) | 0 | 1 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 3 | 6 | 1
RASH (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
FLUSHING (Vascular disorders) | 0 | 1 | 1
HYPOTENSION (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.